CLINICAL TRIAL: NCT02062216
Title: Role of the Inflammatory Receptors in the Pathogenesis of Atherosclerosis
Acronym: Receptors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Other Study IDs: 81/2014/D
Record Dates: First submitted 2014-02-09; First posted 2014-02-13 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Percutaneous coronary intervention; Inflammatory receptors
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI: Patients with ST-elevation myocardial infarction (STEMI) with angiographic evidence of massive thrombosis in the culprit artery undergoing primary percutaneous coronary intervention (PCI)
- STABLE ANGINA: Patients with coronary artery disease in stable conditions scheduled to undergo elective percutaneous coronary intervention and patients with Class I indication to elective percutaneous coronary intervention

SUMMARY:
The primary objective of this study is to assess whether inflammatory receptors play a role in the pathogenesis of atherosclerosis.

DETAILED DESCRIPTION:
Atherosclerosis is a chronic inflammatory disease characterized by lipid deposition and macrophages/foam cell accumulation beneath the arterial intima. Immune competent cells are abundant in atherosclerotic lesions, where they produce mainly proinflammatory cytokines. Macrophages play a central role in each stage of the pathogenesis of atherosclerosis. At the beginning, the so-called foam cells contribute to the formation of early lesions; in mature plaques, macrophages constitute 50% of the cells in the lesion; finally, they are involved in the mechanisms leading to plaque rupture.

The primary objective of this study is to assess whether the inflammatory receptors play a role in the pathogenesis of atherosclerosis.

ELIGIBILITY:
Study Population 1 Patients with ST-elevation myocardial infarction (STEMI) with angiographic evidence of massive thrombosis in the culprit artery undergoing primary percutaneous coronary intervention (PCI)

Criteria

Inclusion Criteria:

* ST-elevation myocardial infarction
* Angiographic evidence of massive thrombosis in the culprit artery
* Indication to primary percutaneous coronary intervention (PCI)
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Study Population 2 Patients with coronary artery disease in stable conditions scheduled to undergo elective percutaneous coronary intervention and patients with

Criteria

Inclusion Criteria:

* A de novo native coronary artery lesions (reference vessel diameter:2.5-3.75 mm)
* Class I indication to elective percutaneous coronary intervention
* Stable conditions and no recent acute coronary syndromes
* Normal baseline values of markers of myocardial damage (creatine kinase, creatine kinase-MB, myoglobin, and troponin I)
* Able to understand and willing to sign the informed CF

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population 1 Patients with ST-elevation myocardial infarction (STEMI) with angiographic evidence of massive thrombosis in the culprit artery undergoing primary percutaneous coronary intervention (PCI)
  Study Population 2 Patients with coronary artery disease in stable conditions scheduled to undergo elective percutaneous coronary intervention and patients with Class I indication to elective percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Level of the inflammatory receptors | Baseline
  Determination of plasmatic level of the inflammatory receptors

SECONDARY OUTCOMES:
C-reactive protein (CPR) | Up to 24 hours after PCI
  Changes 24 hours after PCI in C-reactive protein (CPR)
Fibrinogen | Up to 24 hours after PCI
  Changes 24 hours after PCI in fibrinogen
Plasminogen activator inhibitor (PAI-1) | Up to 24 hours after PCI
  Changes 24 hours after PCI in Plasminogen activator inhibitor (PAI-1)